CLINICAL TRIAL: NCT06846684
Title: A Phase 1, Open-label, Fixed-sequence, Drug-drug Interaction Study to Investigate the Effect of Single and Multiple Oral Doses of SB17170 on the Pharmacokinetics of SB_MDZ in Healthy Adult Subjects
Brief Title: A Open-label, Drug-Drug Interaction With SB_MDZ in Healty Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SPARK Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SMARTT-003
Record Dates: First submitted 2025-02-19; First posted 2025-02-26 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Drug Drug Interaction (DDI)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SB17170 + SB_MDZ (Experimental)
  Interventions: Drug: SB17170; Drug: SB_MDZ

INTERVENTIONS:
Drug: SB17170 — PO, QD
Drug: SB_MDZ — IV

SUMMARY:
This clinical trial is a phase 1, open-label, fixed-sequence, drug-drug interaction study to investigate the effect of single and multiple oral doses of SB17170 on the pharmacokinetics of SB_MDZ in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult subjects aged 19 to 50 years at the time of written consent.
2. Individuals with a body weight of ≥ 50.0 kg, and a Body Mass Index(BMI) of ≥ 18.0 kg/m2 and < 30.0 kg/m2 at the time of screening ☞ BMI(kg/m2) = weight(kg) / {height(m)}2
3. Individuals who have voluntarily provided written consent to participate in the trial, after being fully informed about the study and agreeing to follow all precautions associated with participation.

Exclusion Criteria:

1. Individuals with a clinically significant disease or history in hepatobiliary, renal, nervous, respiratory, immune, hemato-oncology, cardiovascular, urinary system, or psychiatric disorder
2. Individuals with a history of a gastrointestinal disorders (gastrointestinal ulcers, gastritis, stomach cramps, gastroesophageal reflux disease, Crohn's disease, etc) or surgeries (except for simple appendectomy or hernia surgery) that may affect the safety and pharmacokinetic assessment of the investigational product (IP)
3. Individuals with hypersensitivity or significant history of hypersensitivity to drugs, including ingredients of the IP (SB17170 or its metabolite SB1703, SB_MDZ, and benzodiazepine-class drugs) or other drugs (e.g., aspirin, antibiotics)
4. Individuals with a current or historical condition that may increase risk, as determined by the investigator or as indicated in SB_MDZ's product information
5. Individuals who exhibited one or more of the following results in clinical laboratory tests during the screening, including additional tests

   * AST (SGOT), ALT (SGPT) > 60 IU/L
   * Estimated glomerular filtration rate (eGFR, CKD-EPI equation): < 60 mL/min/1.73m2
   * Individuals with a positive result on serology tests (heapatitis B, hepatitis C, human immunodeficiency virus (HIV) and syphilis tests)

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2025-03-27 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Cmax of SB_MDZ | Day 0, 6, 15
AUC of SB_MDZ | Day 0, 6, 15

SECONDARY OUTCOMES:
Tmax of SB_MDZ | Day 0, 6, 15
AUCinf of SB_MDZ | Day 0, 6, 15
T1/s of SB_MDZ | Day 0, 6, 15
CL of SB_MDZ | Day 0, 6, 15
Vz of SB_MDZ | Day 0, 6, 15

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No